CLINICAL TRIAL: NCT03629444
Title: Assessment of Sarcopenia in Patients With Liver Cirrhosis and Its Prognostic Value in Liver Transplant Candidates
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: marwa abdElRazek Ahmed sala.a makhlof (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, marwa abdElRazek Ahmed sala.a makhlof, principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutU2018
Record Dates: First submitted 2018-07-22; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Sarcopenia in Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: ct scan — all patients will be subjected to CT scan and anthroprometric measurments

SUMMARY:
Sarcopenia is a syndrome characterized by progressive and generalized loss of skeletal muscle mass and strength, shown to be prevalent in adults with cancer and common chronic comorbidities such as liver cirrhosis.

The EWGSOP identified a grading for Sarcopenia into pre-sarcopenia (decreased muscle mass with normal strength and physical performance), sarcopenia (decreased muscle mass with decreased strength or performance), severe Sarcopenia (decreased muscle mass, strength and performance) .

Sarcopenia has emerged as an independent predictor of poor prognosis in a variety of clinical conditions.Sarcopenia is clinically important because it can affectthe quality of life of patients with cirrhosis .

Skeletal muscle mass is not only a good indicator of nutrition in patients with cirrhosis, but also has recently been shown to be closely associated with survival prognosis and postoperative complications inHCC.

Combination of sarcopenia and the Model for End-stage Liver Disease (MELD) has been shown to be an excellent model for predicting prognosis in decompensated liver cirrhosis .

Most patients awaiting liver transplantation (LT) are more or less in a state of sarcopenia. Several studies have reported that sarcopenia was associated with worse prognosis.In addition, sarcopenia may be associated with a higher risk of post-transplant infection .

Assessment of sarcopenia in patients with liver cirrhosis:_ The European Working Group on Sarcopenia in Older People recommended that the definition of sarcopenia include not only low muscle mass but also low muscle function . They recommended cutoff values for muscle mass measurements (7.26 kg/m2 for men and 5.5 kg/m2 for women using dual X-ray absorptiometry, and 8.87 kg/m2 for men and 6.42 kg/m2 for women using bioimpedance analysis, handgrip strength (<30 kg for men and <20 kg for women), and usual gait speed (<0.8 m/s).

Aim of the study

* To evaluate sarcopenia in different stages of liver cirrhosis by different diagnostic methods.
* To identify the prognostic value of CT in the diagnosis of sarcopenia .
* To identify effect of sarcopenia inliver transplant candidate.

Patients and methods:

Type of the study:the study is divided into two parts First part: observational descriptive cross sectional study. Second part: follow up of liver transplant candidate group (pre and post liver transplantation) Duration of study: expected duration of the study will be 1.5 years . The 1st part will include all patients admitted to the department for 1 year fulfill inclusion criteria .

2nd part will be 6 ms follow up after liver transplantation. Study population

1. st part : Patients with liver cirrhosis will be evaluated for the presence of sarcopenia.
2. nd part:

   * 13 cases of liver cirrhosis already done liver transplantation in AL Rajhiuneversitiy hospital(which data already recoreded) and any cirrhotic pts will be prerared for liver transplantion within six months.
   * Methods At the study entry, all candidates will be subjected to the following parameters (and 3 month after LT for liver transplant candidates only)
   * Clinical history
   * Clinical examination
   * Abdominal ultrasound
   * Laboratory investigation:

     * Liver function tests
     * Complete blood picture,
     * Kidney function tests,
     * Serum glucose, serum Na+ and K+
     * Hepatitis markers (HBsAg, HCV-Ab)
   * Calculate:

     = Child Pugh score (Pugh et al., 1973) and MELD (Wiesner et al., 2003) scores for assessment ofliver cirrhosis.
   * Anthropometric measurements:

     * Triceps skin fold thickness (TSF) .
     * Measure mid-arm circumference (MAC).
     * Body mass index
     * Hand grip to assess muscle strength
     * Gait speed to assess physical performance
   * Assessment of sarcopenia using CT scan:
   * Assessment of sarcopenia using ultrasound:
   * Assessment of sarcopenia using bioimpedance analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis.
* Age: 18 - 65 years.

Exclusion Criteria:

Cirrhotic patients with:

* Activecomorbid disease e.g. Diabetes mellitus, pulmonary, renal disease (especially .hepatorenal syndrome).
* Malignancy
* Receiving anabolic steroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First part: total coverage of all elligable patients admitted to the department for 1 year who expected 300 patients with liver cirrhosis (only 50 patients will be done CT abdomen due to financial obstacle).
  - Second part:13 cases of liver cirrhosis already done liver transplantation in AL Rajhiuneversitiy hospital and any cirrhotic pts will be prerared for liver transplantion within six months.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
grading of sarcopenia in liver cirrhosis . | about one and half year
  all patients will done CT abdomen with lower limit 38 in female and 53 in male which mean sarcopenia all patients wiill be measure height in cm by stadiometer . all pateints will measure weight in kilograms by weight measuring device. all pateints will be calculated BMI which mean weight\(height)2. with normal range 18.5 to 24.9